CLINICAL TRIAL: NCT06387524
Title: Effects of Eccentric Exercises on Gait Parameters in Patellofemoral Pain Syndrome: A Quasi-Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/1
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Quasi experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): There will be only one group in the study. After application of Mc Connell taping, patients will perform eccentric exercises taught by the therapist for 6 weeks. Mentioned below are detailed protocols for the treatment of patellofemoral pain syndrome.
  Interventions: Procedure: McConnell Taping; Procedure: ECCENTRIC EXERCISES:

INTERVENTIONS:
Procedure: McConnell Taping — Begin with the patient in supine lying with the knee slightly bent. The knee should be completely relaxed and a foam roller or rolled up towel under the knee. Start the tape in line with the middle of the knee cap at the outer aspect of the knee. Using your thumb on top of the sports tape, gently push the patella towards the inner aspect of the knee whilst simultaneously using your fingers to pull the skin at the inner aspect of the knee towards the patella. Finish this taping technique at the inner aspect of the knee ensuring you have created some wrinkling of the skin at the inner aspect of the knee.
Procedure: ECCENTRIC EXERCISES: — Performed for 6 weeks, in 3 sets of 10-12 repetitions each day. Detailed protocol is as under:
  Warm up phase (5 minutes) It will comprise of following components 5 minutes warm up exercise protocol: Marching in place while swinging your arm, rotating toe touching, walking jacks, leg swings, arm circles, shoulder shrugs Eccentric exercises: Each of the following exercise will be performed for 30 seconds, repetitions and hold time will increase with increasing weeks according to patient's stamina.
  Straight leg raise, side lying hip abduction, single leg bridging, supported double leg squatting, hip hikes,supported single leg squatting Following is the detailed description of Cool down phase: Hip stretch, cat cow stretch, oblique stretch, lower back stretch, calf stretch, cross body shoulder stretch

SUMMARY:
This study is a quasi experimental and the purpose of this study is to determine the effects of eccentric exercises on gait parameters in patellofemoral pain syndrome: a quasi - experimental study

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of eccentric exercises on gait parameters in patellofemoral syndrome : a - quasi experimental study

Pain , gait parameters, ROM and dynamic knee valgus angle of young adults (age : 18-35 years ) will be determined using:

1. Numeric pain rating scale
2. Goniometer
3. 30 meter walk test
4. dynamic knee valgus angle via kinovea software Data will be before and after the intervention protocol for each participant. Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Females
* Having pain from at least 2 months
* Pain score greater than 3 on NPRS
* Retro patellar pain in at least two of the following activities:

  1. Ascending, descending stairs
  2. Hooping / jumping
  3. Prolonged sitting with flexed knees
  4. Kneeling and squatting
* Pain on palpation of medial or lateral patellar facet.
* Pain on palpation on anterior portion of medial or lateral femoral condyles.

Exclusion Criteria:

* Diagnosed with Chondromalacia patellae
* Instability of tibiofemoral joint
* Subluxation of patellofemoral joint
* Patellar instability
* Previous surgery of lower limb
* Negative findings on examination of knee ligaments, menisci and bursa.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Dynamic knee valgus angle | 6 weeks
  2D analysis using a video camera will be used to analyze dynamic knee valgus, specifically the inward movement of the knees during task performance. Participants will be instructed to perform a single-leg squat task. They will also be directed to adequately flex the contralateral knee to prevent the foot from touching the floor. A digital video camera positioned at a 90-degree angle to the frontal plane will be placed on a tripod stand 2m in front of the participant's landing point at knee level for 2D video recording purposes. The recorded video will be processed into slow motion and exported to Kinovea software. Dynamic knee valgus angle (DKVA) will be calculated at the intersection point of two lines: the first line connecting markers placed on the anterior superior iliac spine (ASIS) and the middle of the tibio femoral joint, and the second line connecting the middle of the tibio femoral joint and the middle of the ankle mortise.
Hip Range of Motion | 6 weeks
  It will be measured with goniometer
Knee Range of Motion | 6 weeks
  It will be measured with goniometer
Pain intensity | 6 weeks
  Numeric pain rating scale will be used to access pain of the subject pre and post intervention.
Gait Speed | 6 weeks
  Gait speed is the distance that the patient has covered per unit time Calculated as: Gait speed = Distance (m) x time (s)
Cadence | 6 weeks
  Cadence is the number of steps patient takes per unit time. Calculated as: Cadence (steps/min) = steps counted x 60 / time (s)
Stride length | 6 weeks
  Stride length is the distance between two heel strikes of the same foot. Calculated as: SL (m) = speed (m/s) x cycle time (s)
Step length | 6 weeks
  Step length is the vertical distance between heels of two feet. Calculated as: Step length (m) = stride length/2
Cycle length | 6 weeks
  Cycle length is the time between the two heel strikes of one foot. Calculated as: Cycle time (s) = time (s) x 2/steps counted

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan